CLINICAL TRIAL: NCT03261206
Title: Stopping Aminosalicylate Therapy in Inactive Crohn's Disease (STATIC) Study: A Randomized, Open-label, Non-inferiority Trial
Brief Title: Stopping Aminosalicylate Therapy in Inactive Crohn's Disease
Acronym: STATIC
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alimentiv Inc. (Other)
Collaborators: Academic Medical Organization of Southwestern Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RP1610
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Crohn Disease; Remission
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-ASA Continuation (No Intervention): Half of the subjects will continue on aminosalicylate therapy using the same dose and brand for the duration of the study
- 5-ASA Withdrawal (Experimental): Half of the subjects will discontinue their aminosalicylate therapy
  Interventions: Other: 5-ASA Withdrawal

INTERVENTIONS:
Other: 5-ASA Withdrawal — Withdrawal of 5-ASA therapy
  Arms: 5-ASA Withdrawal

SUMMARY:
The purpose of this study is to assess whether withdrawal of aminosalicylate (5-ASA) is non-inferior to continuation of 5-ASA therapy in Crohn's disease (CD) subjects in remission.

DETAILED DESCRIPTION:
Aminosalicylate (5-ASA) agents have proven effective for inducing and maintaining remission in mild to moderate ulcerative colitis (UC) and thus are commonly used as first-line agents for patients with Crohn's disease (CD) in remission. However, there is uncertainty regarding their effectiveness for CD.

In this open-label, randomized study, participants with CD in remission will be allocated to either continue their 5-ASA therapy or withdraw their 5-ASA. The purpose is to investigate if withdrawal of 5-ASA therapy is not unacceptably less effective than continuing on 5-ASA in maintaining CD remission over a 24 month period.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of CD at least 3 months prior to enrollment
* Taking any brand or dosage of an oral aminosalicylate for at least 6 months
* Subject-confirmed compliance with current aminosalicylate therapy (taking at least 75% of prescribed doses)
* CD currently in clinical remission
* Able to participate fully in all aspects of the clinical trial
* Written informed consent obtained and documented

Exclusion Criteria:

* A current diagnosis of UC, indeterminate colitis, microscopic colitis, or diverticular disease-associated colitis
* A diagnosis of short-bowel syndrome
* Active perianal disease
* Active fistulizing disease
* A flare of CD within 3 months prior to enrollment requiring initiation/escalation of medical therapy or surgery
* Use of systemic corticosteroids for CD (2 continuous weeks or more) within 3 months prior to enrollment
* Any major resective bowel surgery for CD (ileal resection, ileocecal resection, proctocolectomy, colectomy, enterectomy, ostomy formation and repair, anastomosis/reanastomosis) within 6 months prior to enrollment
* Unwillingness to stop taking aminosalicylates for the duration of the trial
* Untreated bile salt malabsorption that, in the opinion of the investigator, may interfere with accurate study HBI assessment
* Serious underlying disease other than CD that, in the opinion of the investigator, may interfere with the subject's ability to participate fully in the study
* History of active alcohol or drug abuse that, in the opinion of the investigator, may interfere with the subject's ability to comply with the study procedures
* Currently participating in another interventional trial, or previous participation within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
CD-related complications at 2 years | 24 months
  CD-related complications include either a CD-related or CD treatment-related surgery, hospitalization, or other complication

SECONDARY OUTCOMES:
CD-related complications at 1 year | 12 months
  CD-related complications include either a CD-related or CD treatment-related surgery, hospitalization, or other complication
CD-related or CD-treatment related surgeries at 1 year | 12 months
CD-related or CD-treatment related surgeries at 2 years | 24 months
CD-related or CD-treatment related hospitalizations at 1 year | 12 months
CD-related or CD-treatment related hospitalizations at 2 years | 24 months
Other CD-related or CD-treatment related complications at 1 year | 12 months
  Other complication excludes surgeries or hospitalizations
Other CD-related or CD-treatment related complications at 2 years | 24 months
  Other complication excludes surgeries or hospitalizations
Proportion of patients who require the use of systemic corticosteroids for treatment of CD flares at 1 year | 12 months
Proportion of patients who require the use of systemic corticosteroids for treatment of CD flares at 2 years | 24 months
Time to first CD-related complication | up to 24 months
  CD-related complications include either a CD-related or CD treatment-related surgery, hospitalization, or other complication
Change in disease activity at 6 months | 6 months
  Disease activity assessed by HBI score
Change in disease activity at 12 months | 12 months
  Disease activity assessed by HBI score
Change in disease activity at 24 months | 24 months
  Disease activity assessed by HBI score
Change in self-assessed quality of life at 6 months | Base line and 6 months
  Quality of life assessed with the Crohn's and Ulcerative Colitis Questionnaire 32-item
Change in self-assessed quality of life at 1 year | Base line and 12 months
  Quality of life assessed with the Crohn's and Ulcerative Colitis Questionnaire 32-item
Change in self-assessed quality of life at 2 years | Base line and 24 months
  Quality of life assessed with the Crohn's and Ulcerative Colitis Questionnaire 32-item
Change in C-reactive protein concentration at 6 months | Base line and 6 months
Change in C-reactive protein concentration at 1 year | Base line and 12 months
Change in C-reactive protein concentration at 2 years | Base line and 24 months
Change in fecal calprotectin concentration at 1 year | Base line and 12 months
Change in fecal calprotectin concentration at 2 years | Base line and 24 months
Change in CD-related drug treatment costs at 2 years | 12 months prior to enrollment and 24 months after enrollment
  Estimated drug treatment costs before and after enrollment
Change in CD-related and total healthcare costs at 2 years | 12 months prior to enrollment and 24 months after enrollment
  Estimated costs before and after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Vipul Jairath, MD, Principal Investigator — Western University; London Health Sciences Centre; Gordon Moran, MD, Principal Investigator — University of Nottingham
Locations (46):
- Canada (12):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Dr. Jesse Siffledeen Professional Medical Corporation, Edmonton, Alberta
  - (G.I.R.I.) GI Research Institute, Vancouver, British Columbia
  - Discovery Clinical Services Ltd., Victoria, British Columbia
  - University of Manitoba - Health Sciences Centre, Winnipeg, Manitoba
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Scott Shulman Medical Professional Corporation, North Bay, Ontario
  - Taunton Surgical Center, Oshawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Dr. O. Tarabain Medicine Professional Corporation, Windsor, Ontario
  - McGill University Healthcare, Montreal, Quebec
- Italy (8):
  - IRCCS Policlinico San Donato, San Donato Milanese, Milan Italy
  - Ospedale San Raffaele S.r.I., Milan, Milan
  - UOC Gastroenterologic UOS Malattie Infiammatorie Intestinali, Ospedali, Roma, Rome
  - IRCCS De Bellis, Castellana Grotte, Via Turi
  - Luigi Vanvitelli of Campania, Catania
  - Intituto Clinico Humanitas, Milan
  - Azienda Ospedale-Universita Padova, Padua
  - Campus Bio-Medico University of Rome, Roma
- Ukraine (4):
  - BYK - Kyiv, Kyiv
  - Danylo Halytsky Lviv National Medical University, Lviv
  - Odesa Regional Clinical Hospital, Odesa
  - Ternopil University Hospital, Ternopil
- United Kingdom (22):
  - Warrington and Halton Hospitals NHS Foundation Trust, Warrington, Cheshire
  - Darlington Memorial Hospital, Darlington, Durham
  - Basildon and Thurrock University Hospitals NHS Foundation Trust, Basildon, Essex
  - Royal Blackburn Hospital, Blackburn, Lancashire
  - St. Marks Hospital, Harrow, Middlesex
  - Sherwood Forest Hospitals NHS Foundation Trust - Kings Mill Hospital, Sutton in Ashfield, Nottinghamshire
  - Barnsley Hospital NHS Trust, Barnsley, Yorkshire
  - Bedford Hospital NHS Trust, Bedford
  - Southmead Hospital, North Bristol NHS Trust, Bristol
  - Northern Care Alliance NHS Group - Fairfield General Hospital, Bury
  - West Suffolk Hospital, Bury St Edmunds
  - ESNEFT Colchester Gen Hospital, Colchester
  - Dudley Group NHS Foundation Trust, Dudley
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - University Hospitals of Leicester NHS Trust - Leicester Royal Infirmary, Leicester
  - Royal Free Hospital, London
  - Guy's and St. Thomas' Hospitals NHS Trust, London
  - Luton and Dustable Hospital Foundation Trust, Luton
  - Nottingham University Hospitals NHS Trust and University of Nottingham, Nottingham
  - Royal Berkshire NHS Foundation Trust, Reading
  - Salford Ryal NHS Foundation Trust, Salford
  - Airedale NHS Foundation Trust, Steeton

IPD SHARING:
Plan to Share IPD: No